CLINICAL TRIAL: NCT04621435
Title: Imaging of Solid Tumors Using FAP-2286
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Thomas Hope (Other)
Collaborators: Society of Abdominal Radiology (Other)
Responsible Party: Sponsor-Investigator, Thomas Hope, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20929; NCI-2020-11728 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumors, Adult; Metastatic Cancer
Keywords: PET; 68Ga-FAP-2286; 64Cu-FAP-2286
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CLOSED - 68Ga-Dosimetry population (Cohort 1a) (Experimental): PET imaging will begin 30 +/-10 minutes, 60 +/-15 minutes and 120 +/-20 minutes after injection of 68Ga-FAP-2286. Contrast may be administered if clinically indicated.
  Interventions: Drug: Gallium-68 labelled (68Ga-) FAP-2286; Procedure: Positron Emission Tomography (PET) imaging
- CLOSED - 64Cu-Dosimetry population (Cohort 1b) (Experimental): PET imaging will begin 60±15 minutes, 240±30 minutes after injection, and a second PET imaging will be performed 24±2 hours after initial injection of 64Cu-FAP-2286. Contrast may be administered if clinically indicated.
  Interventions: Procedure: Positron Emission Tomography (PET) imaging; Drug: Copper-64 labeled (64Cu-) FAP-2286
- Participants with metastatic disease (Cohort 2) (Experimental): Participants with metastatic disease will have PET imaging 50-100 minutes after injection of 68Ga- or 64Cu- FAP-2286. Contrast may be administered if clinically indicated.
  Interventions: Drug: Gallium-68 labelled (68Ga-) FAP-2286; Procedure: Positron Emission Tomography (PET) imaging; Drug: Copper-64 labeled (64Cu-) FAP-2286
- Participants without metastatic disease (Cohort 3) (Experimental): Participants without metastatic disease will have PET imaging 50-100 minutes after injection of 68Ga- or 64Cu- FAP-2286. Contrast may be administered if if clinically indicated.
  Interventions: Drug: Gallium-68 labelled (68Ga-) FAP-2286; Procedure: Positron Emission Tomography (PET) imaging; Drug: Copper-64 labeled (64Cu-) FAP-2286

INTERVENTIONS:
Drug: Gallium-68 labelled (68Ga-) FAP-2286 — The dose will be 3 to 8 millicurie (mCi) +/- 10% given intravenously at a single time prior to imaging
  Other Names: 68Ga-FAP-2286
  Arms: CLOSED - 68Ga-Dosimetry population (Cohort 1a); Participants with metastatic disease (Cohort 2); Participants without metastatic disease (Cohort 3)
Procedure: Positron Emission Tomography (PET) imaging — Participants will be scanned for approximately 30 to 45 minutes
  Other Names: PET
Drug: Copper-64 labeled (64Cu-) FAP-2286 — The dose will be 3.5 to 5.5 millicurie (mCi) +/- 10% given intravenously at a single time prior to imaging
  Other Names: 64Cu-FAP-2286
  Arms: CLOSED - 64Cu-Dosimetry population (Cohort 1b); Participants with metastatic disease (Cohort 2); Participants without metastatic disease (Cohort 3)

SUMMARY:
This is a multi-arm prospective trial that evaluates the ability of a novel imaging radiolabeled agents to detect metastatic cancer in participants with solid tumors using a gallium 68 (68Ga-) or copper 64 (64Cu-) FAP-2286 tracer. FAP-2286 is a peptidomimetic molecule that that binds to Fibroblast Activation Protein (FAP). FAP is a transmembrane protein expressed on cancer-associated fibroblasts, and has been shown to be present on a number of solid tumors.

DETAILED DESCRIPTION:
Initially the investigator(s) will focus on imaging breast, pancreas, sarcoma, prostate cancer, bladder cancer, colon cancer, and head and neck cancer.

STUDY AIMS

1. Determine the dosimetry for gallium-68 labelled (68Ga-) and 64Cu- FAP-2286.
2. Evaluate the uptake and retention of radiotracer in a variety of solid tumors with FAP-2286.
3. Evaluate the ability of FAP-2286 to detect metastatic disease.

PRIMARY OBJECTIVES

1. All cohorts: Safety of 68Ga- and 64Cu-FAP-2286.
2. Cohort 1a: determine the organ dosimetry of 68Ga-FAP-2286.
3. Cohort 1b: determine the organ dosimetry of 64Cu-FAP-2286.
4. Cohort 2: To assess the feasibility of detecting tumor uptake using FAP-2286.
5. Cohort 3: To determine the feasibility of detecting metastatic disease using FAP-2286.

EXPLORATORY OBJECTIVES

1. To detect the sensitivity of FAP-2286 PET compared to conventional imaging for the detection of metastatic disease, and when available sensitivity compared to Fluorodeoxyglucose (FDG) PET (FDG-PET).
2. Correlation of FAP-2286 uptake with FAP expression determined by immunohistochemistry.
3. Compare biodistribution of 68Ga-FAP-2286 and 64Cu-FAP-2286 in normal organs and blood pool based on renal function.
4. Determine impact of administered dose of FAP-2286 on image quality.
5. Compare the feasibility of detecting tumor uptake using 68Ga-FAP-2286 and 64Cu-FAP-2286

A repeat radiolabeled FAP-2286 PET may be obtained after initiation of subsequent treatment in order to evaluate changes in PET uptake due to treatment effect. Participants will be followed through the day of the last injection of radiolabeled FAP-2286 for evaluation of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years.
2. Histopathologically confirmed solid tumors in one of the following cohorts:

   a. Cohort 1 (n=11): measurable disease is not required for this cohort.

   i. Agnostic to tumor type.

   b. Cohort 2 (n=95): Metastatic disease present on conventional imaging defined as having RECIST 1.1 measurable disease or multiple bone metastases. Note: Presence of absence of metastatic disease for eligibility determination will be assessed by reviewing medical records. Screening imaging will not be conducted for this study.

   i. Pathologically confirmed breast cancer, pancreatic adenocarcinoma, sarcoma, castrate-resistant prostate cancer, bladder cancer, or colon cancer.

   ii. Pathologically confirmed cancer other than noted above (basket subgroup, n=10).

   c. Cohort 3 (n=85): No evidence of metastatic disease as defined as the absence of RECIST 1.1 measurable disease or bone metastases. Note: Presence of absence of metastatic disease for eligibility determination will be assessed by reviewing medical records. Screening imaging will not be conducted for this study.

   i. Participants can be imaged at initial staging with what is judged by the treating physician to be high risk disease and where the presence of metastatic disease would greatly impact treatment planning and prognosis. Participants may also be imaged after definitive therapy (surgery, chemotherapy or radiation therapy) if in the determination of the treating physician or investigator there is a high risk of disease recurrence that would also impact treatment plan and/or prognosis.

   ii. Pathologically confirmed head and neck cancer or bladder cancer.
3. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Unlikely to comply with protocol procedures, restrictions and requirements and judged by the Investigator to be unsuitable for participation.
2. Known pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Estimated)
Dates: Start 2020-12-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Count of participants with treatment-emergent adverse events | Until end of day on the day of the injection (1 day total)
  The frequency and severity of treatment emergent adverse events following FAP-2286 injection will be descriptively reported as classified and graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0
Proportion of radiation-absorbed doses of radiolabeled FAP-2286 (Cohorts 1a/1b only) | Up to 3 days
  Volumes of interest of 68Ga- and 64Cu- will be drawn around regions identified on the scans, including the liver, spleen, kidneys, urinary bladder, the central sacrum (for hematopoietic marrow) and whole body. Data will be fitted using the Simulation, Analysis, and Modeling Software II (SAAM II) software. Time integrals of activity will be entered into the Organ Level INternal Dose Assessment/EXponential Modeling (OLINDA/EXM) software, using the reference adult model. The results from all patients enrolled will be combined to allow the calculation of mean, standard deviation (SD), and range of radiation-absorbed doses to individual organs
Standardized Uptake Values (SUVs) (Cohort 2 only) | Up to 3 days
  The maximum Standardized Uptake Value (SUVmax) will be calculated for up to five lesions in each patient, with mediastinal blood pool being used as background activity.
Tumor-to-background (TBR) Ratio (Cohort 2 only) | Up to 3 days
  TBR ratios will be calculated for up to five lesions in each patient, with mediastinal blood pool being used as background activity. The median and range of the measured TBRs will be reported across all RECIST measurable lesions as a table broken down by location (organ metastases, nodal metastases and bone metastases).
Proportion of positive lesions on FAP-2286 PET (Cohort 3 only) | Up to 3 days
  Conventional imaging or CT portion of PET/CT scan will be reviewed in conjunction with the FAP-2286 PET images. Lesions will be characterized as positive on FAP-2286 PET if uptake is greater than 1.5 times higher than mediastinal blood pool and uptake cannot be attributed to physiologic or inflammatory reasons. Conventional imaging or CT portion of PET/CT scan will be interpreted as positive by each lesion if the short axis dimension of lymph nodes is greater than 1 centimeter (cm), and organ metastases measure greater than 1 cm in long axis. The gold standard will be the combination of conventional imaging and FAP-2286 PET in combination with clinical follow-up and histopathology (if available). The number of lesions detected by each modality will be compared and sensitivity will be computed. Since this is a proof-of-concept study, it is not powered for the test of agreement. Nevertheless, the agreement will be tested using McNemar's test.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hope, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No